CLINICAL TRIAL: NCT01858584
Title: Prospective, Comparative, Randomized, Controlled Trial on the Efficacy of the Treatment of Gastroesophageal Reflux Infant With Magnesium Alginate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Dario Ummarino, Doctor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STDMG2013
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Gastroesophageal Reflux; Regurgitation; Vomiting; Chronic Cough
Keywords: GER; Alginate; Regurgitation; questionnaire
MeSH Terms: conditions — Gastroesophageal Reflux; Vomiting; Chronic Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Gastrotuss (Experimental): Gastrotuss baby: syrup based on alginate consisting of: magnesium alginate, simethicone, fructose, xanthan gum, honey, D-panthenol, fluid extracts of Althaea officinalis, Papaver rhoeas, zinc oxide, sodium bicarbonate, sodium hydroxide, p-hydroxybenzoate of methyl-sodium, sodium propyl p-hydroxybenzoate, natural flavors, erythrosine (E127), purified water.
  dosage:
  * Infants weighing <5 kg in 2.5 ml 5-10 min after feeding. In case of regurgitation after administration, 1 ml additional
  * Infants weighing> 5 kg per 5 ml dose after the meal and the evening before putting the baby to sleep The administration should be maximum 3 times per day
  Interventions: Drug: Gastrotuss
- Thickened Formula (Active Comparator): Milk thickened (formulat AR): contains a special thickener derived from corn starch waxy, that maintains its fluidity into the bottle and thickens just inside the stomach of the child, and this makes it easy to use in breastfeeding , as it is usable with a common teat.
  Interventions: Dietary Supplement: thickened milk
- control group (No Intervention)

INTERVENTIONS:
Drug: Gastrotuss — Gastrotuss baby: syrup based on alginate consisting of: magnesium alginate, simethicone, fructose, xanthan gum, honey, D-panthenol, fluid extracts of Althaea officinalis, Papaver rhoeas, zinc oxide, sodium bicarbonate, sodium hydroxide, p-hydroxybenzoate of methyl-sodium, sodium propyl p-hydroxybenzoate, natural flavors, erythrosine (E127), purified water.
  dosage:
  * Infants weighing <5 kg in 2.5 ml 5-10 min after feeding. In case of regurgitation after administration, 1 ml additional
  * Infants weighing> 5 kg per 5 ml dose after the meal and the evening before putting the baby to sleep The administration should be maximum 3 times per day
  Arms: Gastrotuss
Dietary Supplement: thickened milk — Milk thickened (formulat AR): contains a special thickener derived from corn starch waxy, that maintains its fluidity into the bottle and thickens just inside the stomach of the child, and this makes it easy to use in breastfeeding , as it is usable with a common teat.
  Arms: Thickened Formula

SUMMARY:
The results on the efficacy of the formulations based on alginic acid are controversial. Corvaglia et al demonstrated a significant reduction in reflux episodes in preterm infants by evaluation with pH-impedance analysis. This study concludes that the use of alginic acid reduces the acidity of the gastroesophageal reflux (GER) and has a non-systemic effect and a lesser presence of side effects compared to the use of H2-receptor antagonist(H2RA) and proton pump inhibitor (PPI).

DETAILED DESCRIPTION:
Primary outcomes This prospective, randomized, controlled trial aims to determine, in a population of infants within one year of life, suffering from gastroesophageal reflux (GER) the effectiveness of magnesium alginate. The clinical improvement of the patient will be evaluated based on the negativity of the symptom score (4.3.1), assessed using a validated questionnaire on symptoms of GER (I-GERQ Annex A).

Secondary outcomes To compare the efficacy of Magnesium Alginate on GER in infants compared with those of thickened feeding and reassurance, basing on questionnaire results.

ELIGIBILITY:
Inclusion Criteria:

* Age < 1 year
* Suggestive symptoms of gastroesophageal reflux (I-GERQ score > 7)
* Absence of clinical evidence of allergy to cow milk protein or other allergic disorder
* No previous intake of thickened formulas, acid suppressants or drugs
* All parents or guardians must sign a document of informed consent
* Patients affected by chronic disease
* Patients affected by hepatic or renal diseases
* Patients affected by cardiac diseases

Exclusion Criteria:

* Patients affected by chronic disease
* Patients affected by hepatic or renal diseases
* Patients affected by cardiac diseases
* Inability or unwillingness to give informed consent
* Patients wth severe neurologic disease
* Patients affected by cow milk protein allergy
* Previous or ongoing intake of thickened formulas, acid suppressants or drugs

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
efficacy on GER | 2 months
  This prospective, randomized, controlled trial aims to determine, in a population of infants within one year of life, suffering from RGE the effectiveness of magnesium alginate. The clinical improvement of the patient will be evaluated based on the negativity of the symptom score (4.3.1), assessed using a validated questionnaire on symptoms of GER (I-GERQ Annex A).

SECONDARY OUTCOMES:
comparison of treatments | 2 months
  • To compare the efficacy of Magnesium Alginate on GER in infants compared with those of thickened feeding and reassurance.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Staiano, Principal Investigator — Federico II University
Locations (1):
- university of Naples Federico II, Naples, Italy

REFERENCES:
- [Derived] Ummarino D, Miele E, Martinelli M, Scarpato E, Crocetto F, Sciorio E, Staiano A. Effect of magnesium alginate plus simethicone on gastroesophageal reflux in infants. J Pediatr Gastroenterol Nutr. 2015 Feb;60(2):230-5. doi: 10.1097/MPG.0000000000000521. PMID 25079477